CLINICAL TRIAL: NCT02643134
Title: External Physical Vibration Lithecbole Contrast With the Traditional Row of Stone Effect After ESWL: A Multi-center Prospective Randomized Controlled Trial
Brief Title: External Physical Vibration Lithecbole Versus Traditional Row of Stone After Extracorporeal Shockwave Lithotripsy(ESWL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice President of the Hospital, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRER(53)2015
Record Dates: First submitted 2015-12-04; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-08

CONDITIONS: Renal Calculi
Keywords: ESWL; EPVL; PDI(Percussion,Diuresis,Inversion); Randomized Controlled Trial(RCT)
MeSH Terms: conditions — Kidney Calculi | interventions — Lithotripsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): Patients in Group 1 undergo extracorporeal shockwave lithotripsy(ESWL).
  Interventions: Procedure: extracorporeal shockwave lithotripsy
- Group 2 (Other): Patients in Group 2 undergo external physical vibration lithecbole for the treatment after extracorporeal shockwave lithotripsy(ESWL).A multi-dimensional physical harmonic vibration inertial guidance technology
  Interventions: Device: External Physical Vibration Lithecbole

INTERVENTIONS:
Procedure: extracorporeal shockwave lithotripsy — Patients in Group 1 undergo extracorporeal shockwave lithotripsy(ESWL).
  Arms: Group 1
Device: External Physical Vibration Lithecbole — Multi-dimensional physical harmonic vibration inertial guidance technology
  Other Names: Friend-I External Physical Vibration Lithecbole
  Arms: Group 2

SUMMARY:
The traditional stone row method comprises increasing exercise, drink lots of water, drug row of stone and stone row position. External physical vibration lithecbole(EPVL) is a non-invasive device active row of stone, the researchers hope that through this test prospective clinical study to evaluate the effectiveness of in vitro physical vibration row of stones after extracorporeal shockwave lithotripsy(ESWL) treatment of stones discharged, thereby improving after ESWL stone clearance rate.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of external physical vibration lithecbole(EPVL) for the treatment after ESWL treatment of stones discharged，thereby improving after extracorporeal shockwave lithotripsy(ESWL) stone clearance rate. Investigators will do a multi-centers randomized controlled trial(RCT)，and investigators plan to perform this study in 10 hospitals，which are the First Affiliated Hospital of Guangzhou Medical University of China, Department of Urology, The Second Affiliated Hospital of Zhengzhou University of China, Jiangsu Province Hospital, Hubei Province Hospital, Zhongshan Hospital, Tongji Hospital,Hubei provincial people's Hospital,Guilin 181 Hospital，the People' Hospital of Huzhou，The People' Hospital of Shaoyang.

Investigators plan to beginning their study August 2015 and end at July 2016. One hundred and eighty patients with ESWL postoperative residual stone will be enrolled in this study. By simple random sampling technique, all the patients will be assigned to the segment of natural stone row group or physical row of stone group, compared two groups of patients with stone clearance rate and complications, Investigators hope that through this test, improve stone clearance rate after ESWL.

Number:

180cases(90 cases in control group, 90 cases in EPVL group)

Grouping methods:

In this trial, investigators will use equilibrium randomization methods that generate random numerical code table, according to the table, patients are randomly assigned to different groups.

Evaluating indicator Stone-free rate in 4 weeks after ESWL. Incidence rate of complications and adverse reactions after EPVL(fever, hematuria, etc).

Trial method:

Examination before ESWL: blood routine, urine routine, renal function(Cre,BUN), coagulation function; intravenous pyelography(IVP) or CT (radiolucent calculus).

ESWL

Record: duration, frequency, voltage, times.

Method of control group(group1):

ESWL without EPVL; Reexamined by abdominal plain film(KUB) or CT (radiolucent calculus) right after ESWL;

After leaving hospital(without drugs), patients should follow the measures bellowed:

1. the amount of fluid intake is more than 2000ml/d
2. increase physical activity
3. rest in position on uninjured side, patients with lower renal calyx calculus need to invert body.

Method of EPVL group(group2):

Start the treatment of EPVL: the amount of fluid intake is about 1000-2000ml, start the treatment of EPVL when patent's bladder is filling; Reexamined by abdominal plain film(KUB) or CT(radiolucent calculus) right after EPVL;

Record: patients' date, treatment procedure and outcome;

After leaving hospital(without drugs), patients should follow the measures bellowed:

1. the amount of fluid intake is more than 2000ml/d
2. increase physical activity
3. rest in position on uninjured side, patients with lower renal calyx calculus need to invert body;

Follow up timing: return hospital respectively in 1,2 and 4 weeks after EPVL.

Follow up project Laboratory testing: routine urinalysis; Imaging examination: KUB or kidney CT scan (radiolucent calculus) Complications and adverse reactions. Data gathering Fill in follow up table data; Radiological images; IVP or kidney CT scan before ESWL; Reexamined by KUB (radiopaque calculus) or CT (radiolucent calculus) right after EPVL. If stones have been eliminated completely in patients with radiolucent calculus before or at the fourth week of follow-up, investigators must provide kidney CT scan.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-65 years;
2. The diameter of calculus is less than or equal to 15mm;
3. Renal or upper ureteral calculus;
4. There's no urinary tract obstruction below stones, and stones didn't cause complete urinary tract obstruction;
5. Stones are fragmented successfully on single session of ESWL, and the diameter of any of fragments is less than 6mm;
6. Normal renal function,

Exclusion Criteria:

1. Couldn't tolerate EPVL;
2. Urinary tract anomalies, stricture or obstruction;
3. Calculus in diverticulum;
4. Severe hydronephosis;
5. Combined with acute urinary tract infection;
6. Coagulation abnormalities;
7. Morbid obesity(BMI>35kg/m2);
8. Patients with ureteral stent;
9. Stones aren't fragment successfully, or the diameter of at least one fragment is more than 6mm ;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Stone free rate (SFR) | return hospital respectively in 1,2 and 4 weeks after ESWL
  Primary SFR is assessed by abdominal plain film （KUB）at 1,2,4 weeks after ESWL. Stone-free status are defined as either the absence of any residual stone fragments.

SECONDARY OUTCOMES:
extracorporeal physical vibration complications | return hospital respectively in 1,2 and 4 weeks after ESWL
  Complication is defined as any adverse event occurred

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, PH.D and M.D, Study Chair — The First Affiliated Hospital of Guangzhou Medical
Locations (1):
- Department of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China